CLINICAL TRIAL: NCT00152100
Title: Transplantation of Highly Purified Haploidentical CD133 Hematopoietic Cells in Children With Severe Combined Immunodeficiency Syndrome
Brief Title: Transplantation of Hematopoietic Cells in Children With Severe Combined Immunodeficiency Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSCID
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Severe combined immunodeficiency; Transplantation; Haploidentical
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Stem Cell Transplantation; Filgrastim; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stem cell transplant
Drug: Filgrastim, Alemtuzumab
Device: Miltenyi CliniMACS

SUMMARY:
Treatment for severe combined immunodeficiency (SCID) is a medical emergency. A stem cell transplant (immature blood cells that can make other blood cells) from a (MSD) matched sibling donor (brother or sister who is a "match" for your child's immune (HLA) type), usually results in complete correction of immune function. However, most patients lack a matched sibling donor, requiring the use of an alternate donor source.

Transplantation of cells from haploidentical family donors (typically parents) has resulted in immune system correction in the majority of SCID individuals. However, only 65-80% of patients survive greater than one year after this procedure. Failure results from life-threatening infections, graft versus host disease (GvHD) or post-transplant treatment-related effects. Also, for patients that survive beyond one year, B-cell (type of blood cell that fights infection) and natural killer cell function (cell that attacks infections and cancer cells) frequently fail to work, resulting in the need for long-term treatment with intravenous gamma-globulin (IVIg).

In this study, in an effort to restore the overall cell function in patients with SCID, researchers will use a highly purified CD133+ hematopoietic cell graft (stem cell transplant without many mature donor white cells, called T-cells) obtained via use of the Miltenyi CliniMACS device, a device not FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed severe combined immunodeficiency
* Two years of age or younger
* A suitable matched sibling donor is not available

Exclusion Criteria:

* An available matched sibling donor or a confirmed matched unrelated donor
* Patients with DiGeorge syndrome, Zap70, MHC Class II deficiency, or cartilage-hair hypoplasia
* Patients with a Lansky performance score of less than 10, evidence of HIV or a congenital rubella infection or a documented neoplasm
* Patients in whom it is not possible to perform a peripheral blood cell harvest on a haploidentical family member

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2004-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To investigate safety issues related to use of haploidentical highly purified CD133+ hematopoietic cells in patients with SCID
To study the effects (good and bad) of this procedure
To learn if this procedure will result in normal immune function in children with SCID

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kasow, DO, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org